CLINICAL TRIAL: NCT03105895
Title: Multicenter Study on Prevention of Incisional Hernia After Laparotomy With an Onlay Mesh Visible on MRI
Brief Title: Prevention of Incisional Hernia With an Onlay Mesh Visible on MRI
Acronym: VISIBLE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Henares University Hospital (Other)
Collaborators: CARDIOLINK (Unknown)
Responsible Party: Principal Investigator, Miguel A ngel Garci-a Urena, Professor of Surgery, Henares University Hospital
Other Study IDs: HH 02
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Incisional Hernia
Keywords: Incisional hernia; Mesh prevention; Mesh augmentation
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mesh group — An onlay PDVF mesh will be placed as abdominal wall reinforcement

SUMMARY:
It has been demonstrated that incisional hernia incidence after laparotomy can be safely reduced with the addition of a mesh to the conventional closure of the abdominal wall. There still some debate about which is the best position to place this mesh: onlay or sublay. In Europe we have now meshes with CEE approval to be used as reinforcement of abdominal wall closure. The investigators have planned to include 200 patients in a multi center study using an onlay PDVF mesh that can be tracked by magnetic resonance. The patients included will be patients with risk factors for the development of an incisional hernia. The incidence of incisional hernia will be assessed clinically and radiologically after 1 and 2 years follow-up. The incidence of surgical sites occurrences and pain will be also assessed.

ELIGIBILITY:
Inclusion Criteria: Any known risk factor for development of incisional hernia

* > 60 years
* BMI > 30
* DM
* Chronic bronquitis
* Smoking
* Neoplasia
* Renal failure
* Liver failure
* Immnusupression
* Urgent operation

Exclusion Criteria:

* Previous supraumbilical midline laparotomy
* Previous incisional hernia
* Emergency surgery
* Life expectancy of less than 12 months
* Patient´s rejection to participate
* Unable to understand and participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing midline laparotomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Incisional Hernia | 24 months
  Development of an incisional hernia diagnosed clinically or radiologically

SECONDARY OUTCOMES:
Surgical site infection | 30 days
  Wound infection according to CDC guidelines
Surgical site seroma | 30 days
  Seroma ocurrence in the wound
Surgical site hematoma | 30 days
  Hematoma occurrence in the wound
Mesh exposition | 30 days
  Mesh that can be seen during postoperative recovery without skin covarage
Evisceration | 30 days
  Postoperative wound dehiscence
Systemic complications | 30 days
  Any systemic complication occurred in the postoperative period
Chronic mesh infection | up to 2 years postoperative
  Mesh chronically infected that need removal to solve
Abdominal wall pain | Up to 2 years
  VAS score in the follow-up
Length of mesh at MRI 6 weeks | 6 weeks
  Length of the mesh calculated at the MRI planned at 6 weeks
Width of mesh at MRI 6 weeks | 6 weeks
  Width of the mesh calculated at the MRI planned at 6 weeks
Length of mesh at MRI 1 year | 1 year
  Length of the mesh calculated at the MRI planned at 1 year
Width of mesh at MRI 1 year | 1 year
  Width of the mesh calculated at the MRI planned at 1 year

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Puerto Real University Hospital, Puerto Real, Cádiz
  - Sureste Hospital, Arganda, Madrid
  - San Agustín University Hospital, Avilés, Principality of Asturias
  - University Central Hospital of Asturias, Oviedo, Principality of Asturias
  - Nuestra Señora del Prado University Hospital, Talavera de la Reina, Toledo
  - Puerta de Hierro University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Yes
This is study to watch the behavior of an onlay mesh for incisional hernia prevention after laparotomy

REFERENCES:
- [Derived] Rodicio Miravalles JL, Mendez CSM, Lopez-Monclus J, Moreno Gijon M, Lopez Quindos P, Amoza Pais S, Lopez Lopez A, Garcia Bear I, Menendez de Llano Ortega R, Diez Perez de Las Vacas MI, Garcia-Urena MA. Short-term outcomes of a multicentre prospective study using a "visible" polyvinylidene fluoride onlay mesh for the prevention of midline incisional hernia. Langenbecks Arch Surg. 2024 Apr 23;409(1):136. doi: 10.1007/s00423-024-03307-x. PMID 38652308